CLINICAL TRIAL: NCT01592487
Title: Effects of a Breakfast and Snack on Cognitive Function in Preadolescents
Status: Withdrawn | Type: Observational
Why Stopped: Study never started, and there are no plans to initiate.
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 114663
Record Dates: First submitted 2012-05-03; First posted 2012-05-07 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-02

CONDITIONS: Brain Function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Lean BMI: BMI in the 25th - 75th percentile
- Overweight BMI: BMI in the 85th - 95th percentile

SUMMARY:
This study is designed to test how breakfast affects brain function, memory and learning in healthy children.

Hypotheses: Based on the results of our initial study and the relevant literature, it is hypothesized that arousal, attention, and performance will be:

1. Greater in those who eat breakfast relative to those who do not;
2. Greater in lean than in overweight children receiving the higher protein breakfast;
3. Greater in fasting lean than fasting overweight children; and
4. Improved following a morning snack in all study groups.
5. Poorer in children with higher stress-related measures (e.g., higher cortisol levels).
6. Heart rate will be lower in fasting relative to fed participants, and across groups will be higher in overweight children.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* attending 4th or 5th grade
* lean BMI or overweight BMI
* right hand dominance
* no food allergies
* eat breakfast at least 4 mornings/week
* no medications for chronic illness/disorder that may affect outcome (as determined by the PI)

Exclusion Criteria:

* food allergies
* medications that could affect the outcome
* left hand dominance

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: healthy 4th and 5th graders
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States